CLINICAL TRIAL: NCT03128684
Title: The Effects of Lentil-containing Food Products on Satiety and Food Intake in Healthy Adults
Brief Title: The Effects of Lentil-containing Food Products on Satiety and Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government); Saskatchewan Pulse Growers (Other); Pulse Canada (Other)
Responsible Party: Principal Investigator, Alison Duncan, Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: REB16-12-883
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Appetite; Satiety; Food Intake
Keywords: lentils; satiety; appetite; food intake; 24-hour energy intake

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Small Green Lentil Muffin (Experimental)
  Interventions: Other: Small Green Lentil Muffin
- Split Red Lentil Muffin (Experimental)
  Interventions: Other: Split Red Lentil Muffin
- Wheat Muffin (Placebo Comparator)
  Interventions: Other: Wheat Muffin
- Small Green Lentil Chili (Experimental)
  Interventions: Other: Small Green Lentil Chili
- Split Red Lentil Chili (Experimental)
  Interventions: Other: Split Red Lentil Chili
- Rice Chili (Placebo Comparator)
  Interventions: Other: Rice Chili

INTERVENTIONS:
Other: Small Green Lentil Muffin — Consumption of small green lentil muffin; consumption of ad libitum pizza test meal after 180 minutes
  Arms: Small Green Lentil Muffin
Other: Split Red Lentil Muffin — Consumption of split red lentil muffin; consumption of ad libitum pizza test meal after 180 minutes
  Arms: Split Red Lentil Muffin
Other: Wheat Muffin — Consumption of wheat muffin; consumption of ad libitum pizza test meal after 180 minutes
  Arms: Wheat Muffin
Other: Small Green Lentil Chili — Consumption of small green lentil chili; consumption of ad libitum pizza test meal after 180 minutes
  Arms: Small Green Lentil Chili
Other: Split Red Lentil Chili — Consumption of split red lentil chili; consumption of ad libitum pizza test meal after 180 minutes
  Arms: Split Red Lentil Chili
Other: Rice Chili — Consumption of rice chili; consumption of ad libitum pizza test meal after 180 minutes
  Arms: Rice Chili

SUMMARY:
The Lentil Satiety study will examine the effects of replacing wheat and rice with two types of lentils within food products (muffins and chilies) on satiety and food intake in healthy adults.

DETAILED DESCRIPTION:
The Lentil Satiety study will examine the effects of replacing wheat and rice with two types of lentils (small green Eston and red split) within food products (muffins and chilies) on satiety and food intake in healthy adults, for a total of 6 study treatments. A total of 3 to 6 study visits (corresponding to consuming all muffins and/or all chilies) will take place where participants will consume one of the study treatments and subsequently complete satiety questionnaires over 180 minutes to measure satiety as subjective appetite sensations (hunger, fullness, desire to eat, and prospective food consumption). At 180 minutes, participants will receive ad libitum pizza and bottled water to consume until they are comfortably full for a measure of weighed food intake. At the end of each study visit, participants will be given a food scale and instructed to weigh and record all food and drink consumed for the remainder of the day for a measure of 24-hour energy intake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* Age 18 to 40 years old
* BMI 20-30 kg/m2

Exclusion Criteria:

* Blood pressure greater than 140/90 mmHg
* Major medical condition including a history of AIDS or hepatitis
* Medical or surgical event requiring hospitalization within 3 months of randomization
* Any medication use except stable dose (3 months) of oral contraceptives, blood pressure or statin medications
* Tobacco use
* Probiotic supplement use
* Dietary fibre supplement use
* Natural health products (NHPs) used for glycemic control (all other NHPs are ok, as long as stable for 3 months)
* Pulse consumption greater than 4 servings per week
* Food allergy or non-food life threatening allergy
* Pregnant or breastfeeding
* Alcohol consumption of greater than 14 drinks per week or greater than 4 drinks per sitting
* Recent or intended significant weight loss or gain (greater than 4kg in previous 3 months)
* Elite athletes
* Shift workers
* Breakfast skippers
* Score greater than 11, 9, or 8 on the Three Factor Eating Questionnaire (TFEQ) Cognitive Restraint, Disinhibition, and Hunger scales, respectively
* Dislike of frozen pizza

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-09 (Actual)

PRIMARY OUTCOMES:
Satiety | Acute: 0, 15, 30, 45, 60, 90, 120, 150, and 180 minutes after treatment consumption
  Satiety will be measured using 100mm visual analog scales (VAS) rating appetite sensations of hunger, fullness, desire to eat, and prospective consumption
Food Intake | Acute: 180 minutes following consumption of treatment
  Food intake will be measured as kilocalories using an ad libitum cheese pizza test meal

SECONDARY OUTCOMES:
24-hour Energy Intake | Acute: 24 hours
  24-hour energy intake will be measured by providing electronic food scales to participants to weigh and record all food and drink consumed for the rest of the day after leaving the study visit

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutraceutical Research Unit, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clark SL, Ramdath DD, King BV, O'Connor KE, Aliani M, Hawke A, Duncan AM. Food Type and Lentil Variety Affect Satiety Responses but Not Food Intake in Healthy Adults When Lentils Are Substituted for Commonly Consumed Carbohydrates. J Nutr. 2019 Jul 1;149(7):1180-1188. doi: 10.1093/jn/nxz050. PMID 31152672